CLINICAL TRIAL: NCT02210637
Title: Non Attendance at Scheduled Appointments as a Marker of Visits in the Emergency Department, Hospitalization and Mortality
Brief Title: Non Attendance at Scheduled Appointments as a Marker of Mortality and Hospital Admission
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Diego Hernan Giunta, MD, MD, Hospital Italiano de Buenos Aires
Other Study IDs: 2301
Record Dates: First submitted 2014-06-13; First posted 2014-08-07 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Appointments and Schedules; Outpatient Clinics, Hospital/Economics; Emergency Department; Hospitalization; Mortality
Keywords: Appointments and Schedules; Outpatient Clinics, Hospital/Economics; Emergency Department; Hospitalization; Mortality
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Retrospective Cohort: Retrospective Cohort of scheduled outpatient appointment

SUMMARY:
To evaluate the association of non attendance at scheduled appointments with visits in the emergency department, hospitalizations and mortality during one year follow up.

DETAILED DESCRIPTION:
Nonattendance at scheduled appointments at outpatient clinics is a common problem in general medical practice, representing a significant cost to the health care system, and resulting in disruption of daily work planning.Nonattendance at medical appointments has consequences not only for doctors (as it requires a greater use of resources and time), but also for patients, because there may be deterioration in the quality of care, and dissatisfaction associated with delays in obtaining a new appointment

ELIGIBILITY:
Inclusion Criteria:

* Over 17 years.
* Adults who attended, did not attend a scheduled appointment at the Outpatient care system at the Italian Hospital of Buenos Aires (HIBA)

Exclusion Criteria:

- The refusal to register or to the informed consent process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We included all requested appointments (random consecutive sampling) between 2012 and 2013 (24 month).
Sampling Method: Probability Sample
Enrollment: 177083 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 1 year
  Mortality of all causes retrospective assesment from secondary data bases

SECONDARY OUTCOMES:
All cause unprogrammed consult to the emergency department | 1 year
  First emergency department consults from secondary data base in 1 year retrospective
All cause unprogrammed admissions to hospital | 1 year
  First all cause unprogrammed admissions to hospital

CONTACTS AND LOCATIONS:
Overall Officials: Diego H Giunta, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Buenos Aires F.D., Argentina